CLINICAL TRIAL: NCT05240794
Title: Effects of Therapeutic Mobile Game on Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: Arcade Therapeutics Inc. (Unknown)
Responsible Party: Principal Investigator, Tracy Dennis, Professor, Hunter College of City University of New York
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-0015
Record Dates: First submitted 2022-01-24; First posted 2022-02-15 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Experimental group (Experimental): Participants receive active ABM-01 for the study
  Interventions: Device: ABM-01
- Placebo Control (Placebo Comparator): Participants receive a digital control for the study
  Interventions: Device: Digital Control

INTERVENTIONS:
Device: ABM-01 — Gamified computerized behavioral therapy with therapeutic intervention based on Attention Bias Modification Training (ABMT)
  Arms: Experimental group
Device: Digital Control — Placebo control for ABM-01
  Arms: Placebo Control

SUMMARY:
Participants with Social Anxiety Disorder (SAD) will use a digital therapeutic for 30 days, and will complete assessments measuring a broad range of anxiety and mood-related symptoms, with a focus on SAD symptoms, and metrics of functional impairment during this time. After the treatment period, participants will be followed at 6 month and 12 month after the completion of the study.

DETAILED DESCRIPTION:
This study aims to assess the feasibility and efficacy of the digital therapeutic ABM-01 in adults ages 22-65 with SAD. Participants access ABM-01 on their mobile smart phone and complete treatment over a period of 30 days. Enrolled participants will be randomly assigned to one of two groups (Experimental Group and Placebo Control) and be assessed over five periods of time (Baseline Session, 30-Day Treatment Phase, Post-Treatment Session, 6-Month Follow Up Session, 12-Month Follow Up Session).

Participants will complete the 30-Day Treatment Phase as well as the five assessments remotely. During the treatment period, participants complete assessments social anxiety and generalized anxiety symptoms, as well as safety and medication use questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Adults 22-65 at the time of screening
* Meets DSM-5 diagnostic criteria for Social Anxiety Disorder
* Access to and willingness to use computer equipment/smartphone compatible with the product platform over a functional network for the study duration.
* Currently residing in the United States

Exclusion Criteria:

* Risk of suicide or has attempted suicide within 24 months of the screening visit
* Moderate to severe substance use disorder
* Current co-morbid psychiatric diagnosis including PTSD, Schizophrenia, Bipolar Disorder I or II, Autism Spectrum Disorder, or Borderline Personality Disorder
* Currently pregnant or planning to become pregnant during the treatment period

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
The Liebowitz Social Anxiety Scale (LSAS) | Baseline to Treatment End (30 days)
  A 24-item, self-rated scale to assess social anxiety in situations as well as the level of avoidance of those situations. Each question is rated on a 4-point scale, where 0 = none, 1 = mild, 2 = moderate, and 3 = severe. Greater scores indicate greater symptom severity.

SECONDARY OUTCOMES:
The Liebowitz Social Anxiety Scale (LSAS) | Bi-weekly time point and at the 6 and 12 month follow-ups
  A 24-item, self-rated scale to assess social anxiety in situations as well as the level of avoidance of those situations. Each question is rated on a 4-point scale, where 0 = none, 1 = mild, 2 = moderate, and 3 = severe. Scores above 55 indicate social phobia.
Generalized Anxiety Disorder - 7 (GAD-7) | Bi-weekly time point and at the 6 and 12 month follow-ups
  A 7-item self-report measure to assess symptoms of anxiety. Each question is rated on a 4-point scale, 0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day. Scores range from 0-21, where greater scores indicate greater anxiety symptoms.
Beck Anxiety Inventory (BAI) | Baseline to Treatment End (30 days)
  A 21-Item self-report measure to assess symptoms of anxiety. Each question is rated on a 4-point scale, 0 = not at all, 1 = mildly but it didn't bother me much, 2 = moderately - it wasn't pleasant at times, and 3 = severely, it bothered me a lot. Higher scores indicate more severe anxiety symptoms.
State-Trait Anxiety Scale (STAI) | Baseline to Treatment End (30 days)
  A 40-Item self-report measure to assess symptoms of state and trait anxiety. There are 20 questions for state anxiety and 20 questions assessing trait anxiety. Each question is rate on a 4-point scale, where 1 = not at all, 2 = somewhat, 3 = moderately so, and 4 = very much so. Greater scores indicate more severe anxiety symptoms.
Hamilton Anxiety Rating Scale (HAM-A) | Baseline to Treatment End (30 days)
  A 14-Item self-report measure to assess symptoms of anxiety. Each item is scored on a scale of 0 = not present to 4 = severe, with a total score range of 0-56. Greater scores indicate more severe anxiety symptoms.
Depression, Anxiety, and Stress Scale (DASS-21) | Baseline to Treatment End (30 days)
  A 21-Item anxiety, depression, and stress measure. Consisted of anxiety, depression, and stress sub-scales. Each question is rated on a 4-point scale, where 0 = did not apply to me at all, 1 = applied to me to some degree, or some of the time, 2 = applied to me to a considerable degree or a good part of time, and 3 = applied to me very much or most of the time. Greater scores indicate greater symptom severity. Anxiety subscale only.
Generalized Anxiety Disorder-7 (GAD-7) | Baseline to Treatment End (30 days)
  A 7-item self-report measure to assess symptoms of anxiety. Each question is rated on a 4-point scale, 0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day. Scores range from 0-21, where greater scores indicate greater anxiety symptoms.

OTHER OUTCOMES:
Anxiety Sensitivity Index (ASI-3) | Baseline to Treatment End (30 days)
  A 18-Item self-report measure to assess symptoms of anxiety. Each question is rated on a 5-point scale, where 0 = very little, 1 = a little, 2 = some, 3 = much, and 4 = very much. Greater scores on the scale indicate more severe anxiety symptoms.
Positive and Negative Affect Schedule (PANAS) | Baseline to Treatment End (30 days)
  A 20-Item self-reported assessment of positive (10 items) and negative affect (10 items). Each question is rated on a 5-point scale, where 1 = very slightly or not at all, 2 = a little, 3 = moderately, 4 = quite a bit, and 5 = extremely. Greater scores indicate greater positive or negative affect.
Beck Depression Inventory II (BDI-II) | Baseline to Treatment End (30 days)
  A 21-Item self-report measure to assess symptoms of depression. Each question is rated on a 4-point scale, where greater scores indicate greater depressive symptoms.
Patient Health Questionnaire (PHQ-2) | Baseline to Treatment End (30 days)
  A 2-Item health questionnaire that measures the frequency of depressed mood and anhedonia. Each question is rated on a 4-point scale, where 0 = not at all, 1 = several days, 2 = more than half the days, and 3 = nearly every day. Greater scores indicate more severe symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy A Dennis-Tiwary, PhD, Principal Investigator — City University of New York, School of Public Health
Locations (1):
- Hunter College of the City University of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No